CLINICAL TRIAL: NCT06407518
Title: Effects of Preoperative Oral Mmidazolam on Postoperative Pain in Sleep Disturbance or Anxiety Patients Undergoing Laparoscopic Colorectal Cancer Resection- A Prospective, Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: Preoperative Oral Midazolam to Postoperative Pain Relief in Sleep Disturbance or Anxiety Patients With Colorectal Cancer
Acronym: POMPPR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024ZSLYEC-351
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Preoperative; Sleep Disturbance; Anxiety; Midazolam; Pain, Postoperative
Keywords: preoperative; oral midazolam; sleep disturbance; anxiety; postoperative pain; colorectal cancer
MeSH Terms: conditions — Parasomnias; Anxiety Disorders; Pain, Postoperative; Colorectal Neoplasms | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midazolam oral solution Group (Experimental): The intervention drug is midazolam oral solution at a dose of 7-10mg. The starting dosage is 7mg, with subsequent individual increases of 1mg up to a maximum dose of 10mg if patients do not achieve sleep within 30 minutes of administration. The individual dose wil be consistently maintained at the corresponding level every night until the surgery.
  Interventions: Drug: Midazolam oral solution
- Control Group (Placebo Comparator): Placebo is a solution of midazolam oral solution that looks, tastes, and appears the same as the intervention drug, similar to the experimental group increment method.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Midazolam oral solution — Each individual administers the midazolam oral solution nightly from enrollment to the surgry.
  Other Names: Midazolam oral solution, YICHANG HUMANWELL PHARMACEUTICAL
  Arms: Midazolam oral solution Group
Other: Placebo — Each individual administers placebo solution nightly from enrollment to the surgry.
  Arms: Control Group

SUMMARY:
Previous studies have indicated a high incidence of sleep disturbances and anxiety symptoms in individuals with colorectal cancers prior to undergoing surgery, leading to worsened postoperative pain, slower recovery, and higher risk of chronic pain. The enhancement of sleep quality is intricately linked to reducing stress. Preoperative drugs that combine hypnosis and anti-anxiety have not been studied in colorectal cancer patients. Midazolam oral solution is safe and effective for short-term hypnotic and anti-anxiety effects in clinical preoperative settings. In the current randomized controlled clinical trial, 280 patients experiencing sleep disturbance or anxiety prior to colorectal cancer surgery will receive midazolam solution to assess its potential efficacy in reducing postoperative pain, expediting recovery, and decreasing the likelihood of chronic pain. Additionally, the study aims to explore the potential connections between midazolam administration and reductions in stress and inflammation.

DETAILED DESCRIPTION:
Preoperative sleep disturbance and anxiety worsen postoperative pain for patients undergoing surgeries. Research indicates that a significant proportion of patients, ranging from 8.8% to 79.1%, experience disturbances in sleep or anxiety prior to surgery. These preoperative issues have been shown to have lasting and intricate effects on postoperative pain, fatigue, and depression. Therefore, it is imperative for clinical doctors to promptly identify preoperative sleep disturbances and anxiety in order to offer appropriate support to patients.

Colorectal cancer is the fifth leading cause of death in China, with nearly 40% of patients experiencing insomnia before surgery, consistent with our previous studies. A case-control study demonstrated a protective association between improved sleep quality and relief of postoperative pain in colorectal cancers. Furthermore, individuals undergoing laparoscopic colorectal surgery showed a higher likelihood of experiencing visceral pain compared to somatic pain. Acute visceral pain has the potential to progress into chronic visceral pain, resulting in behavioral manifestations such as anxiety, fear, and depression, which may persist and exacerbate into enduring chronic pain, ultimately impacting the individual's quality of life. Currently, studies have shown that disturbed preoperative sleep has become a significant predictor of both acute and chronic postoperative pain. Therefore, finding effective interventions to promote preoperative sleep is a continuing consideration for clinicians.

Pharmacological intervention is the primary approach for preoperative sleep disturbances or anxiety. Finding appropriate drug is a challenge that needs to be solved in the clinical practice. There is currently a lack of evidence-based medical guidelines regarding pharmacologic interventions for preoperative sleep disturbances and anxiety. Research has indicated that zolpidem can enhance sleep quality in patients prior to surgery, decrease the need for analgesics during the procedure, and alleviate postoperative pain. Nevertheless, there is a demand for agents that possess both short-term hypnotic and anxiolytic properties, whereas zolpidem solely exhibits hypnotic effects. Midazolam, a short-acting benzodiazepine, is often used before anesthesia for its short-term hypnotic and anxiolytic effects. Studies have found that midazolam oral solution is safe and effective for short-term use in clinical pre-surgical settings. There are no studies on using oral midazolam solution to improve sleep and reduce anxiety in colorectal cancer patients before surgery. Our previous research found that a dose of 7.2mg can effectively induce sleep with minimal side effects in 50% patients before surgery.

In summary, the present study intends to carry out a prospective,randomized,double-blind,placebo-controlled clinical study to investigate the hypothesis that preoperative oral midazolam solution could reduce acute postoperative pain, promote early recovery, and reduce the risk of chronic pain in patients with poor sleep or anxiety before colorectal cancer surgery. It is postulated that the potential benefits of preoperative oral midazolam solution may be attributed to decreased stress levels, and lowered inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed of informed consent voluntarily; 2. Native Chinese speaker; 3. Age 18-60 years old, male or female; 4. BMI 18-30 kg/m2; 5. American Society of Anesthesiologists (ASA) grade 1 or 2, New York Heart Association (NYHA) gradeⅠor Ⅱ; 6. Non-emergency laparoscopic colorectal cancer resection; 7. General anesthesia with tracheal intubation; 8. Sleep disturbance (the Insomnia Severity Index,ISI≥15 ) or Anxiety (Generalized Anxiety Disorder scale-7,GAD-7≥10 ) from admission to surgery.

Exclusion Criteria:

* 1. Contraindications for Midazolam Oral Solution (According to the Instruction for Midazolam Oral Solution); 2. High risk of Obstructive Sleep Apnea Symptoms (Total score of STOP-Bang scale ≥3 points); 3. Suspected dementia (Total score of Mini-Mental State Examination (MMSE) according to years of education: 0 year≤19 points; 1~6 years≤22 points; above of 6 years≤26 points); 4. Severe depressive symptom within two weeks (Total score of Patient Health Questionnaire-9 (PHQ-9)≥15); 5. History of Neurological and Psychiatric diseases (According to the electronic medical record system); 6. History of Chronic Obstructive Pulmonary Disease (According to the electronic medical record system); 7. History of Heart Failure (According to the electronic medical record system); 8. Intestinal obstruction(The electronic medical record system records those who currently have any type of intestinal obstruction); 9. Liver and renal insufficiency; 10. Have taken opioids or drugs that act on the central nervous system within one week; 11. Take CYP3A4 isoenzyme inhibitors or inducers within one week (According to the Instruction for Midazolam Oral Solution); 12. Consume any alcoholic beverage within 24 hours; 13. Substance abusers (including alcohol, drugs or addictive substances); 14. Pregnant or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate to severe pain on the first postoperative day | on the first postoperative day for Acute Postoperative Pain
  NRS: Numerical Rating Scale, NRS pain score 0-3 for mild, 4-6 for moderate, 7-10 for severe; Moderate to severe pain: Mean NRS pain score ≥4; Mean NRS pain score: Mean pain is defined as the mean of NRS scores of the severest, lightest, average, and present pain within 24 hours using the Brief Pain Inventory Short version (BPIsf).

SECONDARY OUTCOMES:
Mean NRS pain score | on the first postoperative day for Acute Postoperative Pain
  NRS: Numerical Rating Scale, NRS pain score 0-3 for mild, 4-6 for moderate, 7-10 for severe; Mean NRS pain score: Mean pain is defined as the mean of NRS scores of the severest, lightest, average, and present pain within 24 hours using the Brief Pain Inventory Short version (BPIsf).
Mean NRS pain score | on the second postoperative day for Acute Postoperative Pain
  NRS: Numerical Rating Scale, NRS pain score 0-3 for mild, 4-6 for moderate, 7-10 for severe; Mean NRS pain score: Mean pain is defined as the mean of NRS scores of the severest, lightest, average, and present pain within 24 hours using the Brief Pain Inventory Short version (BPIsf).
Mean NRS pain score | on the third postoperative day for Acute Postoperative Pain
  NRS: Numerical Rating Scale, NRS pain score 0-3 for mild, 4-6 for moderate, 7-10 for severe; Mean NRS pain score: Mean pain is defined as the mean of NRS scores of the severest, lightest, average, and present pain within 24 hours using the Brief Pain Inventory Short version (BPIsf).
Incidence of moderate to severe pain | on the second postoperative day for Acute Postoperative Pain
  NRS: Numerical Rating Scale, NRS pain score 0-3 for mild, 4-6 for moderate, 7-10 for severe; Moderate to severe pain: Mean NRS pain score ≥4; Mean NRS pain score: Mean pain is defined as the mean of NRS scores of the severest, lightest, average, and present pain within 24 hours using the Brief Pain Inventory Short version (BPIsf).
Incidence of moderate to severe pain | on the third postoperative day for Acute Postoperative Pain
  NRS: Numerical Rating Scale, NRS pain score 0-3 for mild, 4-6 for moderate, 7-10 for severe; Moderate to severe pain: Mean NRS pain score ≥4; Mean NRS pain score: Mean pain is defined as the mean of NRS scores of the severest, lightest, average, and present pain within 24 hours using the Brief Pain Inventory Short version (BPIsf).
The number of times analgesics being added | on the first postoperative day for Acute Postoperative Pain
  The number of additional postoperative analgesics, by Patient-Controlled Analgesia or prescribed by doctors
The number of times analgesics being added | on the second postoperative day for Acute Postoperative Pain
  The number of additional postoperative analgesics, by Patient-Controlled Analgesia or prescribed by doctors
The number of times analgesics being added | on the third postoperative day for Acute Postoperative Pain
  The number of additional postoperative analgesics, by Patient-Controlled Analgesia or prescribed by doctors
Total scores of the questionnaire of 15-item Quality of Recovery scale | on the first postoperative day
  QoR-15: 15-item Quality of Recovery scale; QoR-15 is a patient-reported measure, and is used to assess global recovery quality after surgery physiologically and psychologically. QoR-15 contents 15 items, which item is constructed by an 11-point numerical rating scale (for positive items, 0="none of the time"to 10="all of the time"; for negative items the scoring are reversed). The total scores are ranging from 0(extremely poor QoR) to 150 (excellent QoR).
Total scores of the questionnaire of 15-item Quality of Recovery scale | on the second postoperative day
  QoR-15: 15-item Quality of Recovery scale; QoR-15 is a patient-reported measure, and is used to assess global recovery quality after surgery physiologically and psychologically. QoR-15 contents 15 items, which item is constructed by an 11-point numerical rating scale (for positive items, 0="none of the time"to 10="all of the time"; for negative items the scoring are reversed). The total scores are ranging from 0(extremely poor QoR) to 150 (excellent QoR).
Total scores of the questionnaire of 15-item Quality of Recovery scale | on the third postoperative day
  QoR-15: 15-item Quality of Recovery scale; QoR-15 is a patient-reported measure, and is used to assess global recovery quality after surgery physiologically and psychologically. QoR-15 contents 15 items, which item is constructed by an 11-point numerical rating scale (for positive items, 0="none of the time"to 10="all of the time"; for negative items the scoring are reversed). The total scores are ranging from 0(extremely poor QoR) to 150 (excellent QoR).
Requirement for propofol when induction of general anesthesia | on the day of colorectal cancer resection and general anesthesia
  Propofol is titrated for the purpose of achieving general anesthesia prior to colorectal cancer resection. Upon reaching the titration endpoint, indicated by an OAAS sedation score of 0, the dosage of propofol administered (in mg/kg) is documented.
  OAAS：Observer's Assessment Alertness/Sedation scale
Incidence of post-anesthesia care unit (PACU) stays longer than 1 hour | on the day of colorectal cancer resection and general anesthesia
  Following the surgical procedure, the patient is relocated to the Post-Anesthesia Care Unit (PACU). Patients may be transferred to the general ward once their postoperative resuscitation meets established standards. Incidence of PACU stays longer than 1 hour is recorded.
The amount of additional analgesics in PACU | on the day of colorectal cancer resection and general anesthesia
  The quantity of supplementary analgesic medications administered in PACU
Incidence of fever in the first 72 hours after surgery | In the third postoperative day
  The incidence of axillary temperatures above 38℃ within 72 hours post-surgery is recorded.
Length of hospital stay after surgery | Days from operation completion to actual hospital discharge (expected 7 days after surgery)
  Length of hospital stay after surgery：hospital stay time (days) from operation completion to actual hospital discharge
The financial burden in the hospital after surgery | Days from operation completion to actual hospital discharge (expected 7 days after surgery)
  Medical costs from operation completion to actual hospital discharge
Incidence of unplanned reoperations within 30 Days after Surgery | within 30 days after surgery
  Incidence of unplanned reoperations within 30 Days after Surgery
Incidence of unplanned admissions within 30 Days after Surgery | within 30 days after surgery
  Incidence of unplanned admissions within 30 Days after Surgery
Total score of The Brief Pain Inventory at the 30th day after surgery | at the 30th day after surgery for chronic Postoperative Pain
  The Brief Pain Inventory: to survey postoperative chronic pain after surgery
Total score of The Brief Pain Inventory at the 90th day after surgery | at the 90th day after surgery for chronic Postoperative Pain
  The Brief Pain Inventory: to survey postoperative chronic pain after surgery
Total score of SF-36 at the 30th day after surgery | at the 30th day after surgery for postoperative health status
  SF-36: The short form (SF)-36 is an instrument to survey postoperative health status.
Total score of SF-36 at the 90th day after surgery | at the 90th day after surgery for postoperative health status
  SF-36: The short form (SF)-36 is an instrument to survey postoperative health status.
Number of patients still taking pain medication on day 30 after surgery | on the 30th day after surgery
  Number of patients still taking pain medication on day 30 after surgery
Number of patients still taking pain medication on day 90 after surgery | on the 90th day after surgery
  Number of patients still taking pain medication on day 90 after surgery
Incidence of post-traumatic stress disorder (PTSD) at 30 days post-surgery | on the 30th day after surgery
  The prevalence of post-traumatic stress disorder as measured by the PC-PTSD scale at 30 days following surgical procedures.
  PC- PTSD：Primary Care Post traumatic Stress Disorder
Incidence of post-traumatic stress disorder (PTSD) at 90 days post-surgery | on the 90th day after surgery
  The prevalence of post-traumatic stress disorder as measured by the PC-PTSD scale at 90 days following surgical procedures.
  PC- PTSD：Primary Care Post traumatic Stress Disorder
The ratio of neutrophils to lymphocytes in peripheral blood on the first day after surgery | on the first day after surgery
  The ratio of neutrophils to lymphocytes in peripheral blood on the first day after surgery
The ratio of neutrophils to lymphocytes in peripheral blood on the third day after surgery | on the third day after surgery
  The ratio of neutrophils to lymphocytes in peripheral blood on the third day after surgery
The ratio of platelets to lymphocytes in peripheral blood on the first day after surgery | on the first day after surgery
  The ratio of platelets to lymphocytes in peripheral blood on the first day after surgery
The ratio of platelets to lymphocytes in peripheral blood on the third day after surgery | on the third day after surgery
  The ratio of platelets to lymphocytes in peripheral blood on the third day after surgery
C-reactive protein levels in peripheral blood on the first day after surgery | on the first day after surgery
  C-reactive protein levels in peripheral blood on the first day after surgery
C-reactive protein levels in peripheral blood on the third day after surgery | on the third day after surgery
  C-reactive protein levels in peripheral blood on the third day after surgery
Opioid consumption in milligrams of intravenous morphine equivalents within three days after surgery | within three days after surgery
  Opioid consumption in milligrams of intravenous morphine equivalents within three days after surgery
Opioid consumption in milligrams of intravenous or oral morphine equivalents within 30 days after surgery | within 30 days after surgery
  Opioid consumption in milligrams of intravenous or oral morphine equivalents within 30 days after surgery
Opioid consumption in milligrams of intravenous or oral morphine equivalents within 90 days after surgery | within 90 days after surgery
  Opioid consumption in milligrams of intravenous or oral morphine equivalents within 90 days after surgery
Incidence of nausea (requiring treatment) and vomiting within three days after surgery | within three days after surgery
  Incidence of nausea (requiring treatment) and vomiting within three days after surgery
Incidence of patients mobilising on the first day after surgery | on the first day after surgery
  Incidence of patients mobilising on the first day after surgery
time until first flatus after surgery in days | time until first flatus after surgery in days (generally, within the three days after surgery )
  time until first flatus after surgery in days
Incidence of complications related to surgery within 30 days after surgery | within 30 days after surgery
  Incidence of complications related to surgery within 30 days after surgery [ complication grade according to Clavien-Dindo（No complications，Grade I-II，Grade IIIa + IIIb，Grade IV，Grade V）]

OTHER OUTCOMES:
Salivary cortisol | Days from admission to the day of surgery (expected 5 days before surgery)
  preoperative Salivary cortisol
Cytokine group | on the surgery day (before general anesthesia and surgery)
  Peripheral blood being collected before surgery
Endocannabinoids | on the surgery day (before general anesthesia and surgery)
  Peripheral blood being collected before surgery

CONTACTS AND LOCATIONS:
Overall Officials: sanqing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No